CLINICAL TRIAL: NCT02601196
Title: IVF Outcome Following Treatment With Ulipristal Acetate for Myomatous Uterus After at Least One IVF Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eran Zilberberg, Doctor, IVF unit, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-15-2101-EZ-CTIL
Record Dates: First submitted 2015-10-15; First posted 2015-11-10 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Women With Leiomyoma After at Least One Unsuccessful IVF Treatment
Keywords: Leiomyoma; Infertility; IVF; Ulipristal acetate
MeSH Terms: conditions — Leiomyoma; Infertility | interventions — ulipristal acetate

ARMS (1):
- Ulipristal acetate treatment (Other): Women who receive UPA treatment before another IVF cycle.
  Interventions: Drug: Ulipristal acetate

INTERVENTIONS:
Drug: Ulipristal acetate — Transvaginal US and diagnostic hysteroscopy - to ascertain suitability. A therapeutic course of ulipristal acetate 5 mg per day for 13 weeks. After completion of the treatment protocol - another TVUS, diagnostic hysteroscopy and histological examination of the endometrium - to assess results of UPA treatment.
  Another IVF cycle.

SUMMARY:
Hypothesis:

After reviewing the relevant medical data the investigators assume that treating a woman with intramural fibroid not distorting the uterine cavity or mostly intramural with less than 50% submucosal component with Ulipristal Acetate (UPA) for a 13 weeks course would reduce the fibroid size and improve her chance for conceiving by IVF treatment.

Materials & Methods:

Study design: A proof of concept prospective not randomized study. The patients: About 20 women treated in the fertility and IVF unit after at least one IVF failure, with mostly intramural (IM) fibroid [class 2-5 by FIGO (International Federation of Gynecology and Obstetrics) classification system] in the size of >4 cm confirmed by Transvaginal ultrasound (TVUS) and diagnostic hysteroscopy.

After US examination and diagnostic hysteroscopy to ascertain suitability for this study, the investigators will offer a course of 13 weeks treatment with UPA 5 mg per day.

One month after cessation of treatment the investigators will perform another TVUS examination & diagnostic hysteroscopy plus endometrial biopsy in order to assess the endometrial & uterine status and will conduct an additional IVF cycle, using the same stimulation protocol undertaken during the immediate cycle previous to the UPA treatment course.

DETAILED DESCRIPTION:
Ulipristal Acetate - Study design

Introduction:

Leiomyomas are well established factors to affect fertility. The key factor for fertility disturbance is the fibroid location and not its size. The presence of submucosal fibroids has long been known to reduce fertility as opposed to subserosal fibroids which do not alter fertility. The effect of intramural fibroids on fertility is still a mystery.

These findings were best described in a meta-analysis of 23 studies:

* With no respect to location, women with fibroids have a lower chance for ongoing pregnancy or live birth (RR 0.7, 95% CI 0.59-0.83) and a greater chance for spontaneous abortion (RR 1.68, 95% CI 1.37-2.05).
* Women with fibroids that were submucosal or intramural with an intracavitary component were less likely to become pregnant (RR 0.36, 95% CI 0.18-0.74) and more likely to have a spontaneous abortion (RR 1.7, 95% CI 1.4-2.1).
* The picture is less clear for women with intramural fibroids. Overall, studies of women with fibroids that did not distort the uterine cavity were less likely to become pregnant (RR 0.81, 95% CI 0.70-0.94), less likely to have an ongoing pregnancy or to deliver a live newborn (RR 0.7, 95% CI 0.58-0.85) and more likely to have a spontaneous abortion (RR 1.7, 95% CI 1.2-2.5).
* In addition to these findings, women with cavity-distorting fibroids who undergone myomectomy had a significant increase in conception rate (RR 2.03, 95% CI 1.08-3.83).
* There were no significant differences between women who had myomectomy for intramural fibroids and those who did not go through surgical treatment, although the data for this issue is quite lame.

Another strong evidence for the relevance of intramural fibroids for fertility can be found in a meta-analysis that evaluated the association between non-cavity-distorting intramural fibroids and IVF outcome, this study shows a significant decrease in the live birth (RR 0.79, 95% CI 0.70 -0.88) and clinical pregnancy rate (RR 0.85, 95% CI 0.77 - 0.94) in women with non-cavity-distorting intramural fibroids compared with those without fibroids, following IVF treatment.

Ulipristal:

Ulipristal acetate (UPA) is a selective progesterone receptor modulator (SPRM) prescribed for women with symptomatic leiomyomas. Few phase 3 studies were conducted in order to prove its clinical use and efficacy in treating women suffering from fibroids.

* PEARL (PGL4001 Efficacy Assessment in Reduction of Symptoms Due to Uterine Leiomyomas) I was a randomized, double-blind, placebo controlled trial (48 patients in the placebo arm, 95 treated with daily dosage of 5 mg & 94 with 10 mg of UPA) proving that treatment with UPA 5 mg or 10 mg once daily for a 13 weeks course is efficient in controlling uterine bleeding (91% & 92% respectively) in comparison to placebo (19%), P<0.001 for each dose. The rates of amenorrhea were 73%, 82% and 6% respectively. The median change in total fibroid volume was -22%, -12% & +3% (p=0.002 for the 5 mg group & 0.006 for the 10 mg group in comparison to the placebo group).
* PEARL II was a double blind non-inferiority trial comparing UPA (5 mg or 10 mg once daily) treatment for 3 months to once-monthly IM Leuprolide acetate 3.75 mg (97 patients in the 5 mg arm, 103 in the 10 mg arm & 101 treated by Leuprolide acetate). The rates of uterine bleeding were comparable between the three groups - 90%, 98%, 89%. Median times to amenorrhea were 7 days, 5 days, 21 days - respectively. Adverse effects in the matter of moderate to severe hot flashes were much more common for women treated with Leuprolide acetate - 40% in comparison to those treated with UPA (11% for the 5 mg group & 10% for the 10 mg group, p<0.001 for both groups).

In November 2014 Luyckx et al. published a retrospective analysis of a series of 52 patients from one medical center (participants in PEARL II or PEARL III) - of these patients, 21 wished to conceive upon treatment completion - 15 of them (71%) succeeded for a total of 18 pregnancies.

* Median time to conceive was 10 months after completion of therapy.
* Two women who did not need myomectomy after completion of the UPA treatment achieved 3 of the pregnancies.
* 15 pregnancies were after myomectomy (8 by laparoscopy, 7 by laparotomy).
* 6 of the pregnancies (6 of 18, 33%) resulted in early missed abortion while 12 of the pregnancies ended in the live births of 13 babies. The relative high ratio of miscarriage can be related to the age of the women (median 36.4 years) and to high proportion of IVF (3/6 miscarriages).
* Only one of the deliveries was a vaginal delivery, 7 had elective cesarean delivery and 4 had emergent cesarean section.
* There was no significant fibroid regrowth during pregnancy.
* There was only one fetal anomaly in this cohort - in a patient who was treated by a new UPA course while she was already pregnant (unexpectedly) - a fetus showing ectopic right kidney on the inferior pole of the left kidney. A review of pregnancies after exposure to mifepristone to induce abortion or UPA given as emergency contraception shows no additional risk for congenital anomalies.

Selective progesterone receptor modulators as UPA are well known to induce endometrial modification known as PAEC (Progesterone receptor modulators Associated Endometrial Changes) - these changes are benign, non-proliferative & non-physiological. This histological pattern is apparent in a large proportion of women after 13 weeks UPA treatment course (in PEARL I - 74.2% of the patients in the 5 mg group & 70.4% in the 10 mg group; in PEARL II 65.1% in the 5 mg group & 69.8% among the treated with 10 mg UPA). Endometrial biopsies taken six months after treatment cessation showed return to normal histological endometrial appearance. In both RCT's all endometrial biopsy examinations taken after week 13 showed only benign changes except: (a) one patient after 5 mg UPA treatment whose specimen showed simple hyperplasia and (b) one patient in the placebo group with complex atypical hyperplasia.

Hypothesis:

After reviewing the relevant medical data the investigators assume that treating a woman with intramural fibroid not distorting the uterine cavity or mostly intramural with less than 50% submucosal component with UPA for a 13 weeks course would reduce the fibroid size and improve her chance for conceiving by IVF treatment.

Materials & Methods:

Study design: A proof of concept prospective not randomized study. The patients: About 20 women treated in our fertility and IVF unit after at least one IVF failure, with mostly intramural fibroid [class 2-5 by FIGO classification system] in the size of >4 cm confirmed by TVUS and diagnostic hysteroscopy.

After US examination and diagnostic hysteroscopy to ascertain suitability for our study, we will offer a course of 13 weeks treatment with UPA 5 mg per day.

One month after cessation of treatment the investigators will perform another TVUS examination & diagnostic hysteroscopy plus endometrial biopsy in order to assess the endometrial & uterine status and will conduct an additional IVF cycle, using the same stimulation protocol undertaken during the immediate cycle previous to the UPA treatment course.

The data:

Demographic data - Age, BMI. Obstetrical data - Gravida, para. Gynecological data - Hormonal profile, uterus size, fibroids features (location, size), infertility features (duration, cause), past stimulation and IVF treatment variables.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women in the age of 18-44 years
* At least after one failure in IVF treatment
* Normal responders (more than 3 oocytes retrieved in previous controlled ovarian hyperstimulation treatment).
* Intramural fibroid between 4-10 cm, not distorting the uterine cavity

Exclusion Criteria:

* Intolerance for UPA treatment
* Fibroids distorting the uterine cavity
* Poor responder

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy | About 10-12 weeks after embryo transfer
  Number of viable pregnancies at about 10-12 weeks of gestation
Clinical pregnancy | 3 weeks after embryo transfer
  Number of cases with gestational sac per US exam

SECONDARY OUTCOMES:
Uterus size | A month after the end of UPA treatment
  The size of the uterus per TVUS after UPA treatment
Fibroids status | A month after the end of UPA treatment
  Status of fibroids per TVUS after UPA treatment (number, location, volume cm^3)
Number of oocytes retrieved | Right after ovarian pick-up
  Number of oocytes retrieved during ovarian pick-up
Number of embryos | About 3 days after OPU (ovum pick-up)
  Number of developing embryos in the laboratory
Number of top quality embryos | 3 days after OPU
  The number of day 3 embryos with 7-8 cells with less than 15% fragmentation
Live birth | Until 40 weeks past embryo transfer
  Number of pregnancies ended in a live birth

REFERENCES:
- [Background] Klatsky PC, Tran ND, Caughey AB, Fujimoto VY. Fibroids and reproductive outcomes: a systematic literature review from conception to delivery. Am J Obstet Gynecol. 2008 Apr;198(4):357-66. doi: 10.1016/j.ajog.2007.12.039. PMID 18395031
- [Background] Pritts EA, Parker WH, Olive DL. Fibroids and infertility: an updated systematic review of the evidence. Fertil Steril. 2009 Apr;91(4):1215-23. doi: 10.1016/j.fertnstert.2008.01.051. Epub 2008 Mar 12. PMID 18339376
- [Background] Casini ML, Rossi F, Agostini R, Unfer V. Effects of the position of fibroids on fertility. Gynecol Endocrinol. 2006 Feb;22(2):106-9. doi: 10.1080/09513590600604673. PMID 16603437
- [Background] Sunkara SK, Khairy M, El-Toukhy T, Khalaf Y, Coomarasamy A. The effect of intramural fibroids without uterine cavity involvement on the outcome of IVF treatment: a systematic review and meta-analysis. Hum Reprod. 2010 Feb;25(2):418-29. doi: 10.1093/humrep/dep396. Epub 2009 Nov 12. PMID 19910322
- [Background] Donnez J, Tatarchuk TF, Bouchard P, Puscasiu L, Zakharenko NF, Ivanova T, Ugocsai G, Mara M, Jilla MP, Bestel E, Terrill P, Osterloh I, Loumaye E; PEARL I Study Group. Ulipristal acetate versus placebo for fibroid treatment before surgery. N Engl J Med. 2012 Feb 2;366(5):409-20. doi: 10.1056/NEJMoa1103182. PMID 22296075
- [Background] Donnez J, Tomaszewski J, Vazquez F, Bouchard P, Lemieszczuk B, Baro F, Nouri K, Selvaggi L, Sodowski K, Bestel E, Terrill P, Osterloh I, Loumaye E; PEARL II Study Group. Ulipristal acetate versus leuprolide acetate for uterine fibroids. N Engl J Med. 2012 Feb 2;366(5):421-32. doi: 10.1056/NEJMoa1103180. PMID 22296076
- [Background] Luyckx M, Squifflet JL, Jadoul P, Votino R, Dolmans MM, Donnez J. First series of 18 pregnancies after ulipristal acetate treatment for uterine fibroids. Fertil Steril. 2014 Nov;102(5):1404-9. doi: 10.1016/j.fertnstert.2014.07.1253. Epub 2014 Sep 17. PMID 25241376
- [Background] Bernard N, Elefant E, Carlier P, Tebacher M, Barjhoux CE, Bos-Thompson MA, Amar E, Descotes J, Vial T. Continuation of pregnancy after first-trimester exposure to mifepristone: an observational prospective study. BJOG. 2013 Apr;120(5):568-74. doi: 10.1111/1471-0528.12147. Epub 2013 Jan 24. PMID 23346916
- [Background] Gemzell-Danielsson K, Rabe T, Cheng L. Emergency contraception. Gynecol Endocrinol. 2013 Mar;29 Suppl 1:1-14. doi: 10.3109/09513590.2013.774591. PMID 23437846
- [Background] Williams AR, Bergeron C, Barlow DH, Ferenczy A. Endometrial morphology after treatment of uterine fibroids with the selective progesterone receptor modulator, ulipristal acetate. Int J Gynecol Pathol. 2012 Nov;31(6):556-69. doi: 10.1097/PGP.0b013e318251035b. PMID 23018219